CLINICAL TRIAL: NCT03113448
Title: 0.075% Capsaicin Lotion for the Treatment of Painful Diabetic Neuropathy: A Randomized, Double- Blind, Crossover, Placebo-Controlled Trial
Brief Title: 0.075% Capsaicin Lotion for the Treatment of Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Assawin Chomjit, Director, Clinical research, Thammasat University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTU-EC-IM-5-195/59; TCTR20170407001 (Other: Thai Clinical Trials Registry)
Record Dates: First submitted 2017-04-09; First posted 2017-04-13 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Peripheral Diabetic Neuropathy
Keywords: capsaicin; neuropathic pain; diabetic neuropathy; topical lotion
MeSH Terms: conditions — Neuralgia; Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.075% Capsaicin Lotion (Active Comparator): 0.075% Capsaicin Lotion is used for application at skin area involved with symptomatic neuropathic pain (both feet or/and hands), 3-4 times a day, everyday for 8 weeks then stop
  Interventions: Drug: 0.075% Capsaicin Lotion; Drug: placebo
- Placebo Lotion (Placebo Comparator): Placebo Lotion is used for application at skin area involved with symptomatic neuropathic pain (both feet or/and hands), 3-4 times a day, everyday for 8 weeks then stop
  Interventions: Drug: 0.075% Capsaicin Lotion; Drug: placebo

INTERVENTIONS:
Drug: 0.075% Capsaicin Lotion — To apply 3-4 times per day, every day until 8 weeks then stop
Drug: placebo — To apply 3-4 times per day, every day until 8 weeks then stop

SUMMARY:
To study that 0.075% capsaicin lotion is safe, well tolerated and provide significant pain relief in patients with PDN compared with placebo lotion as a randomized, double- Blind, crossover, placebo-controlled trial

DETAILED DESCRIPTION:
Neuropathy is one of the most common complications in both type 1 and type 2 diabetes mellitus. The most common symptom is a symmetrical, chronic, axonal, length-dependent sensorimotor polyneuropathy.

Topical capsaicin formulations are widely used to manage pain. Low-concentration creams, lotions, and patches intended for daily skin application have been available in most countries since the early 1980s.

We study 0.075% capsaicin lotion is safe, well tolerated and provide significant pain relief in patients with PDN compared with placebo lotion as a randomized, double- Blind, crossover, placebo-controlled trial for 20 weeks throughout the study in 42 participants. All participants are provided both 0.075% capsaicin lotion and placebo lotion. Each agent will be applied for 8 weeks then stop for 4 weeks, after that another agent will be used for 8 weeks. We keep following up all of them by calling and appointment to get information in effectiveness and adverse effect at 0,2,4,8,12,14,16,20 week, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. DM type 2 over 1 year
2. Clinical presentation of peripheral sensory such as burning pain
3. DN4 score from 4 points
4. Good consciousness to tell their score with informed consent agreement
5. No adding dosage of previous pain control medications at least 4 weeks
6. HbA1C 6.5-9.0%

Exclusion Criteria:

1. Improper application site of skin for topical drugs such as abrasion wound.
2. Allergic history of Capsaicin
3. No intention to join the study with any reasons
4. Other previous medications used that effect to peripheral neuropathy such as Carboplatin, Cisplatin, Colchicine, Dapsone, Etoposide, Ethambutol, Indomethacin, Isoniazid, Lithium, Metronidazole, Phenytoin, Pyridoxine, Statins, Stavudine (d4T) or conditions worsening peripheral nerves following that poor nutrition, kidney failure, chronic alcoholism, vitamin deficiency, Hypothyroidism

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (0-100 mm.) | 20 week
  scale

SECONDARY OUTCOMES:
Short-form McGill Pain Questionnaire(SF-MPQ) | 20 week
  scale
Neuropathic Pain Scale (NPS) | 20 week
  scale

CONTACTS AND LOCATIONS:
Overall Officials: Kongkiat Kulkantrakorn, Professor, Study Chair — Thammasat University Hospital; Pasiri Sithinamsuwan, Study Director — Phramongkutklao College of Medicine
Locations (1):
- Thammasat University Hospital, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangwani-Mordani S, Goodman CF, Galor A. Novel Treatments for Chronic Ocular Surface Pain. Cornea. 2023 Mar 1;42(3):261-271. doi: 10.1097/ICO.0000000000003193. Epub 2022 Dec 19. PMID 36729473